CLINICAL TRIAL: NCT00304551
Title: A Phase II/III Study of Peginterferon Alfa-2a in Combination With Ribavirin for the Treatment of CHC With Compensated LC
Brief Title: A Study of Peginterferon Alfa-2a in Combination With Ribavirin in Chronic Hepatitis C (CHC) Patients With Compensated Liver Cirrhosis (LC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JV19595
Record Dates: First submitted 2006-03-05; First posted 2006-03-20 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Liver Cirrhosis; Chronic Hepatitis C
Keywords: CHC with compensated LC
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: peginterferon alfa-2a 180μg; Drug: ribavirin
- 2 (Experimental)
  Interventions: Drug: peginterferon alfa-2a 90μg; Drug: ribavirin
- 3 (No Intervention)

INTERVENTIONS:
Drug: peginterferon alfa-2a 180μg — 180μg（s.c.）/week for 48 weeks
  Arms: 1
Drug: peginterferon alfa-2a 90μg — 90μg(s.c.)/week for 48 weeks
  Arms: 2
Drug: ribavirin — 600, 800, or 1,000 mg X 2(p.o.)/day
  Arms: 1; 2

SUMMARY:
This study evaluated the clinical response of the efficacy and safety of the combination therapy of peginterferon alfa-2a and ribavirin, compared with an antiviral treatment-free group in CHC patients with compensated LC.

Additionally, this study evaluated the dosage reactivity and the pharmacokinetic characteristics of the combination therapy of peginterferon alfa-2a and ribavirin in CHC patients with compensated LC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 75 years-old with quantifiable serum HCV-RNA (≥ 500 IU/mL), elevated serum alanine aminotransferase activity (≥ 45 IU per liter) within sixty days of screening, and proven CHC with compensated LC (Child-Pugh A) on liver biopsy.

Exclusion Criteria:

* Patients with neutropenia (fewer than 1,500 neutrophils per cubic millimeter)
* Thrombocytopenia (fewer than 75,000 platelets per cubic millimeter)
* Anemia (less than 12 g hemoglobin per deciliter )
* Hepatitis B co-infection; decompensated liver disease.
* Organ transplant
* Creatinine clearance less than 50 milliliters per minute
* Poorly controlled psychiatric disease
* Poorly controlled diabetes
* Malignant neoplastic disease
* Severe cardiac or chronic pulmonary disease
* Immunologically mediated disease
* Retinopathy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Sustained virological response, defined as undetectable hepatitis C virus (HCV)-RNA (< 50 IU per milliliter [IU/mL]) | week 24 from the end of treatment

SECONDARY OUTCOMES:
Biochemical response (normalization of serum alanine aminotransferase activity) | at the end of treatment and week 24 form the end of treatment
Virological response (HCV-RNA < 50 IU per milliliter) | at the end of treatment and week 24 form the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Takehiko Aoshima, Study Director — Clinical Research Department 4, Chugai Pharmaceutical Co., Ltd.
Locations (8):
- Japan (8):
  - Chugoku, Chugoku
  - Hokkaido Region, Hokkaido
  - Kanto Region, Kanto
  - Kinki Region, Kinki
  - Kyusyu Region, Kyusyu
  - Shikoku Region, Shikoku
  - Tohoku Region, Tōhoku
  - Tokai Region, Tōkai